CLINICAL TRIAL: NCT05070611
Title: Efficacy of Intense Pulsed Light in the Treatment of Recurrent Chalazia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0562
Record Dates: First submitted 2021-09-09; First posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Chalazion
Keywords: Chalazion; IPL; Meibomian gland function
MeSH Terms: conditions — Chalazion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recurrent chalazia with IPL-MGX (Experimental): The patients whose lesions had failed to respond to warm compresses and antibiotic and steroid treatment underwent incision and curettage. One week after lesion incision, the E-Eye machine (E-SWIN company, France) IPL treatment was administered to the skin area below the lower eyelid. After removal of the ultrasound gel, meibomian gland expression (MGX) was performed with forceps-shaped meibomian gland compressor.
  Interventions: Device: IPL-MGX

INTERVENTIONS:
Device: IPL-MGX — One week after lesion incision, the E-Eye machine (E-SWIN company, France) IPL treatment was administered to the skin area below the lower eyelid.13 Before treatment, the eyes were protected with opaque goggles and ultrasound gel was applied on the patient's face from tragus to tragus including the nose to conduct the light.

SUMMARY:
The purpose of the present study was to investigate the efficacy of intense pulse light and meibomian glands expression in cases of recurrent chalazion after surgery.

DETAILED DESCRIPTION:
We hypothesized that IPL application on the skin adjacent to eyelids after chalazion surgery will result in better meibomian gland function and lower recurrence. To date, it has not been previously reported the outcomes of the use of this technology for the management of chalazions recurrence. The purpose of the present study was to investigate the efficacy of intense pulse light and meibomian glands expression in cases of recurrent chalazion after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients had chronic unilateral recurrent chalazia that failed to resolve after conservative treatment that included warm compresses and antibiotic and steroid ophthalmic ointments.

Exclusion Criteria:

* (1) any intraocular inflammation, ocular infection, allergy, ocular surgery, or ocular trauma in the past 6 months; (2) any eyelid diseases or structural abnormality; (3) any systematic diseases may lead to dry eye or MGD; (4) skin cancer or pigmented lesion in the treatment zone.

Ages: 24 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of chalazia | an average of 1 year
  The recurrence rate of the recurrent chalazia

SECONDARY OUTCOMES:
NITBUT | an average of 1 year
  non-invasive tear film breakup time
meibomian expressibility and quality | an average of 1 year
  The expressibility and quality score of the meibum
TMH | an average of 1 year
  tear meniscus height

CONTACTS AND LOCATIONS:
Overall Officials: lin lin, Study Chair — Second Affiliated Hospital of Zhejiang University Hospital
Locations (1):
- Second Affiliated Hospital of Zhejiang University Hospital, Hangzhou, China